CLINICAL TRIAL: NCT05557357
Title: Electroacupuncture With or Without Combined Warm Needling for Tinnitus: Study Protocol for A Randomized, Waitlist-controlled Trial
Brief Title: Electroacupuncture With or Without Combined Warm Needling for Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lai Fun HO, PhD (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor-Investigator, Lai Fun HO, PhD, Chinese Medicine Practitioner I, Pok Oi Hospital
Organization: Pok Oi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EAnEAWN-Tinnitus
Record Dates: First submitted 2022-09-18; First posted 2022-09-28 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Tinnitus; Tinnitus, Subjective
Keywords: Tinnitus; Acupuncture; Moxibustion; Warm Needling; Clinical Trial; Randomized Controlled Trial
MeSH Terms: conditions — Tinnitus | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- EA Group (Experimental): Subjects assigned to EA group will receive EA treatment twice weekly for 5 weeks.
  Interventions: Procedure: Electroacupuncture (EA)
- EAWN Group (Experimental): Subjects assigned to EAWN group will receive EAWN treatment twice weekly for 5 weeks.
  Interventions: Procedure: Electroacupuncture Combined With Warm Needling (EAWN)
- Waitlist Control Group (Other): Subjects assigned to waitlist control group will not receive treatment during the 10-week waiting period after baseline assessment.
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Procedure: Electroacupuncture (EA) — Electroacupuncture (EA) treatment following standardized procedures will be conducted for 2 sessions per week for 5 consecutive weeks. Each session of treatment will last for 25 min.
  The acupoints that will be stimulated are Tinggong (SI19) and Yifeng (TE17) of the affected side, Baihui (GV20) and Yintang (GV24+), bilateral posterior temporal line (MS11), and Zhongzhu (TE3) and Zusanli (ST36) of the affected side.
  For electroacupuncture (EA), electrical stimulation will be applied using an EA apparatus, with pairs of electrodes connecting the needles at ipsilateral SI19 and TE17, GV20 and GV24+, and bilateral MS11.
  Arms: EA Group
Procedure: Electroacupuncture Combined With Warm Needling (EAWN) — Electroacupuncture combined with warm needling (EAWN) treatment following standardized procedures will be conducted for 2 sessions per week for 5 consecutive weeks. Each session of treatment will last for 25 min.
  The acupoints that will be stimulated are SI19 and TE17 (affected side), GV20 and GV24+, bilateral MS11, and TE3 and ST36 (affected side).
  For electroacupuncture (EA), electrical stimulation will be applied using an EA apparatus, with pairs of electrodes connecting the needles at ipsilateral SI19 and TE17, GV20 and GV24+, and bilateral MS11.
  For warm needling (WN), two moxa sticks will be ignited and attached one by one to the needle handle of each acupoint of SI19 and TE17.
  Arms: EAWN Group
Other: Waitlist Control — No treatment will be provided during the 10-week waiting period after baseline assessment.
  Arms: Waitlist Control Group

SUMMARY:
This randomized controlled trial aims to evaluate the efficacy and safety of either electroacupuncture alone or combined with warm needling in reducing tinnitus loudness and improving the impairment caused by tinnitus in Hong Kong.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, assessor-blind, three-arm, parallel-group, randomized waitlist-controlled trial. A total of 90 eligible subjects with tinnitus will be recruited and randomly assigned to electroacupuncture (EA), electroacupuncture combined with warm needling (EAWN) or waitlist control with n=30 subjects each group. The entire study period will last for 10 weeks, including a 5-week intervention period and a 5-week follow-up period. Outcome measures include the loudness of tinnitus and the Tinnitus Handicap Inventory. Any adverse event will be observed and recorded for safety assessment. The study findings will provide evidence to determine the efficacy and safety of electroacupuncture with or without combined warm needling for tinnitus in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with subjective tinnitus;
* Male and female, age 50 to 70 years old;
* Unilateral or bilateral tinnitus for 0.5-24 months;
* Loudness of tinnitus rated 3 points or more on a 0-10 numeric rating scale (NRS) at the time of enrollment; and
* Agree to sign the informed consent form voluntarily.

Exclusion Criteria:

* Known disease conditions that could cause tinnitus such as Meniere's syndrome, acoustic duct diseases, and middle ear diseases;
* History of head trauma;
* Currently using cardiac pacemaker or metal implants;
* Known severe cardiac diseases, cerebrovascular diseases, renal diseases, or hematologic diseases;
* Known severe psychiatric or psychological disorder;
* Pregnant, lactation or expecting a pregnancy during the study period;
* Severe needle phobia;
* Known hypersensitive reaction after acupuncture and moxibustion treatment or an inability to cooperate with the acupuncture and moxibustion procedure;
* Incapable to understand and answer the questions of the assessors in the study; and
* Other factors deemed unsuitable for inclusion in the study by investigators.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Change in Tinnitus Loudness | Baseline, Week 5, and Week 10
  A 0-10 numeric rating scale (NRS) will be used for rating loudness of tinnitus. Higher score indicates greater tinnitus loudness and its influence.

SECONDARY OUTCOMES:
Change in Tinnitus Handicap Inventory (THI) | Baseline, Week 5, and Week 10
  THI is a 25-item self-report measure to determine tinnitus handicap severity with good reliability and validity. The THI total score ranges from 0 to 100, with higher score denoting higher level of severity.

OTHER OUTCOMES:
Adverse Events | Up to 10 weeks
  Any adverse event related to study treatment will be recorded and analyzed throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanqi GUO, Principal Investigator — Pok Oi Hospital
Locations (3):
- China (3):
  - Pok Oi Hospital-Chinese Medicine Polyclinic (Tin Shui Wai), Hong Kong
  - Pok Oi Hospital-The Chinese University of Hong Kong Chinese Medicine Clinic cum Training ad Research Centre (Yuen Long District), Hong Kong
  - Pok Oi Hospital-The Chinese University of Hong Kong Chinese Medicine Clinic cum Training and Research Centre (Shatin District), Hong Kong

IPD SHARING:
Plan to Share IPD: No